CLINICAL TRIAL: NCT00657332
Title: Clinical and Pathologic Studies in Neuroendocrine Tumors
Status: Withdrawn | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: George Albert Fisher M.D. Ph.D., Stanford University School of Medicine
Other Study IDs: IRB-8988; 98132; END0005; NCT00657332
Record Dates: First submitted 2008-04-09; First posted 2008-04-14 (Estimated); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Carcinoid Tumor; Neuroendocrine Tumors
MeSH Terms: conditions — Carcinoid Tumor; Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — biopsy of tumor, blood sample and/or urine samples.

INTERVENTIONS:
Procedure: blood sample draw
Procedure: urine sample

SUMMARY:
This research involves the study of neuroendocrine tumors in order to better understand how the disease grows and spreads. This study requires will use tissue collected from from biopsies performed during your regular medical care (i.e. tissue leftover after your diagnosis has been made) and/or blood and urine samples. This study may lead to the development of special materials that could be used, in the future, to treat neuroendocrine tumors or to follow the response of neuroendocrine tumors to treatment

ELIGIBILITY:
Inclusion Criteria:- Patients are eligible if they have a histologically proven neuroendocrine tumor and are 18 years of age or older

- Ability to understand and the willingness to sign a written informed consent document. Exclusion Criteria:None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: neuroendocrine tumor patients
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2007-07; Primary Completion 2008-06-17 (Estimated); Study Completion 2008-06-17 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: George Albert Fisher M.D. Ph.D., Principal Investigator — Stanford University